CLINICAL TRIAL: NCT04894383
Title: A Study Into the Use of Prefabricated Orthotics in Shoes, in Combination With Using Indoor Comfort Sandals With built-in Arch Support vs. the Sole Use of Prefabricated Orthotics in Shoes Alone, for the Treatment of Plantar Fasciitis. A Randomised Control Trial
Brief Title: Plantar Fasciitis and the Use of Orthotics as Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Talita Cumi Ltd. (Industry)
Collaborators: Aetrex Worldwide Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFPETFETS002
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prefabricated Orthotics in shoes & indoor comfort sandals with built-in arch support (Experimental): Participants from Group A will receive an L400 Compete Orthotic (https://www.aetrex.com/search?q=l420&search-button=&lang=en_US) and an Aetrex comfort sandal with built-in arch support (https://www.aetrex.com/aetrex-flips-black-L3000M.html?lang=en_US or https://www.aetrex.com/fiji-flips-women-watermelon-L7009W.html?lang=en_US) according to participants shoe size. The investigators will send an instruction sheet along with the Orthotic in the post, explaining how to use it. Alternatively, an online video tutorial on how to use the Orthotic will also be available throughout the study. The group will be asked to continue with usual activities, using the orthotic/comfort sandal wherever possible.
  Interventions: Device: Aetrex L420 Compete Orthotic; Device: Aetrex indoor comfort sandal with built-in arch support
- Prefabricated Orthotics in shoes only (Active Comparator): Group B will receive an L400 Compete Orthotic (https://www.aetrex.com/search?q=l420&search-button=&lang=en_US) alone. The investigators will send an instruction sheet along with the Orthotic in the post, explaining how to use it. Alternatively, an online video tutorial on how to use the Orthotic will also be available throughout the study. The group will be asked to continue with usual activities, using the Orthotic wherever possible.
  Interventions: Device: Aetrex L420 Compete Orthotic

INTERVENTIONS:
Device: Aetrex L420 Compete Orthotic — An orthotic insole to be inserted into shoes. Orthotic for low arches to flat feet with no forefoot pain, featuring a posted heel to control over-pronation and provide balance. Features Aetrex Arch Support to help biomechanically align the body & help prevent common foot pain such as Plantar Fasciitis, Arch Pain and Metatarsalgia.
Device: Aetrex indoor comfort sandal with built-in arch support — An indoor comfort sandal with built-in arch support to be used at home. Provides extreme cushioning, shock absorption and durability. Arch support helps to stabilize and align feet and also helps to relieve common foot pain & plantar fasciitis.
  Arms: Prefabricated Orthotics in shoes & indoor comfort sandals with built-in arch support

SUMMARY:
To investigate whether the use of prefabricated Orthotics in shoes, in combination with the use of indoor comfort sandals with built-in arch support, benefits the treatment of plantar fasciitis more than the sole use of prefabricated Orthotics in shoes alone.

DETAILED DESCRIPTION:
The usual symptom of plantar fasciitis is "first-step pain", though plantar heel pain in general can be broadly associated with plantar fasciitis. Although most of the cases resolve within 10 months, 10% develop chronic plantar fasciitis. The pathomechanics of the condition is assumed to be due to excessive tensile loading, exacerbated by abnormal biomechanics of the legs such as pes planus, leg length discrepancy, and tightness of calf muscles.

Foot Orthotics are commonly used in the conservative treatment of plantar fasciitis. It is thought that foot Orthotics reduce the symptoms of plantar fasciitis by reducing strain in the fascia during standing and ambulation. A handful of randomized controlled trials have evaluated the effects of foot Orthotics from a patient's perspective. However, systematic reviews of these trials have concluded that the evidence for the effectiveness of foot Orthotics in the treatment of plantar fasciitis is poor and that further investigation is needed. In addition, the limitation of the success of using orthotics may be because Orthotics can only be used in conjunction with shoes. Many people may not wear shoes when at home, meaning the Orthotics are not being used during this time. The feet are therefore unsupported for a significant number of hours when weight-bearing (walking and standing) without shoes. This research, therefore, involves testing the addition of contoured comfort sandals with built-in arch support that can be worn while at home, as well as the Orthotics which will be worn during the day with shoes. Contemporaneous research on Orthotics is limited to only using Orthotics and there are no studies that use both the Orthotics and comfort sandal.

This is a randomised control trial that will be conducted over a 6-month period, during which participants will be asked to provide data in the form of completed surveys at 5 points throughout the study period. The aim of the study is to investigate whether the use of prefabricated Orthotics in shoes, in combination with the use of indoor comfort sandals with built-in arch support, benefits the treatment of plantar fasciitis more than the sole use of prefabricated Orthotics in shoes alone.

The study population will include 104 participants who will be randomised into a study and control group. Participants in the study group will be asked to insert the Orthotics into normal footwear and to use them wherever possible. Participants will also be instructed to use the comfort sandal with built-in arch support when not using shoes whilst at home. Participants in group B will only be asked to use the Orthotic inserted into daily footwear wherever suitable (i.e. when outside of the home). Participants from both groups will be asked to continue with normal activities throughout the study period.

During the 6 month study period, all participants will be asked to complete and submit surveys at baseline, 3 weeks, 6 weeks, 3 months and 6 months from entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Have been experiencing symptoms of Plantar Fasciitis for at least 2 months. A diagnosis of plantar fasciitis will be made on the criteria that the pain is located on the medial aspect of the heel on palpation and the pain is worst the first thing in the morning.
* Aged 19-75 years old

Exclusion Criteria:

* Prior operations on the foot,
* Prior treatments apart from analgesia in the last 12 months e.g. corticosteroid injections,
* Congenital or acquired foot and ankle abnormalities which prevent the use of normal footwear.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in Pain as assessed by a Visual Analogue Scale (VAS) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  Pain will be collected on via a self-report Visual Analogue Scale (VAS) as follows: 0 to 10 where 0 is 'No Pain' and 10 is 'The worst imaginable pain'.

SECONDARY OUTCOMES:
Changes in Foot health status as assessed by the Foot Health Status Questionnaire (FHSQ) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  Foot Pain & Functionality scores will be collected using the FHSQ or Foot Health Status Questionnaire. The Foot Health Status Questionnaire is designed to assess foot pain, foot health and its relation to quality of life. The questionnaire has four domains consisting of 13 key items. The four domains are; foot pain, foot function, footwear and general foot health. The current study will only use the 2 subsections of Foot Pain and Foot Function. In these subsections, participants will be required to rate foot pain in the last week from 1 (none) to 5 (severe), how often the participant experienced different types of foot pain during the last week from 1 (never) to 5 (always), how much the participants feet interfered with everyday activities in the last week from 1 (not at all) to 5 (extremely) and overall foot health from 1 (excellent) to 5 (poor). Previous research has found the FHSQ to exhibit a strong degree of context, criterion and construct validity with high retest reliability.
Changes in overall health as assessed by The Global Rating Scale of Change (GROC scale) | Baseline, 3 weeks, 6 weeks, 3 months and 6 months
  The Global Rating Scale of Change, or the GROC scale, will be used in the current study to assess participants overall health. This will give further insight into the effectiveness of the interventions. It is an 11 point scale from -5 to + 5. "-5" denotes "very much worse", "0" denotes "unchanged" and "+5" denotes "completely recovered".

CONTACTS AND LOCATIONS:
Overall Officials: George Ampat, MBBS, MS, FRCS, Principal Investigator — Talita Cumi Ltd.
Locations (1):
- Talita Cumi LTD., Southport, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, data will be fully anonymised. Only non-identifiable, anonymised data will be archived along with the publication for use of other researchers. For instance, the age, sex, and study results of participants will be archived indefinitely as a supplementary document to the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available at the completion of the study on 31/12/2022. It will be available for other researchers indefinitely.
Access Criteria: The non-identifiable data will be openly available as a supplementary document to the publication.

REFERENCES:
- [Background] Roos E, Engstrom M, Soderberg B. Foot orthoses for the treatment of plantar fasciitis. Foot Ankle Int. 2006 Aug;27(8):606-11. doi: 10.1177/107110070602700807. PMID 16919213
- [Background] Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. No abstract available. PMID 15152061
- [Background] Wearing SC, Smeathers JE, Urry SR, Hennig EM, Hills AP. The pathomechanics of plantar fasciitis. Sports Med. 2006;36(7):585-611. doi: 10.2165/00007256-200636070-00004. PMID 16796396
- [Background] Bennett PJ, Patterson C. The foot health status questionnaire (FHSQ): a new instrument for measuring outcomes of foot care. Australasian J Podiatr Med. 1998;32:55-9.
- [Background] Bennett PJ, Patterson C, Dunne MP. Health-related quality of life following podiatric surgery. J Am Podiatr Med Assoc. 2001 Apr;91(4):164-73. doi: 10.7547/87507315-91-4-164. PMID 11319246
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Result] Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID 15134610
- [Result] Clement DB, Taunton JE, Smart GW, McNicol KL. A Survey of Overuse Running Injuries. Phys Sportsmed. 1981 May;9(5):47-58. doi: 10.1080/00913847.1981.11711077. PMID 27453020
- [Result] Davis PF, Severud E, Baxter DE. Painful heel syndrome: results of nonoperative treatment. Foot Ankle Int. 1994 Oct;15(10):531-5. doi: 10.1177/107110079401501002. PMID 7834059
- [Result] Kogler GF, Solomonidis SE, Paul JP. Biomechanics of longitudinal arch support mechanisms in foot orthoses and their effect on plantar aponeurosis strain. Clin Biomech (Bristol). 1996 Jul;11(5):243-252. doi: 10.1016/0268-0033(96)00019-8. PMID 11415628
- [Result] Kitaoka HB, Luo ZP, An KN. Analysis of longitudinal arch supports in stabilizing the arch of the foot. Clin Orthop Relat Res. 1997 Aug;(341):250-6. PMID 9269181
- [Result] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Result] Crawford F, Atkins D, Young P, Edwards J. Steroid injection for heel pain: evidence of short-term effectiveness. A randomized controlled trial. Rheumatology (Oxford). 1999 Oct;38(10):974-7. doi: 10.1093/rheumatology/38.10.974. PMID 10534548
- [Result] Acevedo JI, Beskin JL. Complications of plantar fascia rupture associated with corticosteroid injection. Foot Ankle Int. 1998 Feb;19(2):91-7. doi: 10.1177/107110079801900207. PMID 9498581
- [Result] Leach R, Jones R, Silva T. Rupture of the plantar fascia in athletes. J Bone Joint Surg Am. 1978 Jun;60(4):537-9. PMID 27524
- [Result] Anderson RB, Foster MD. Operative treatment of subcalcaneal pain. Foot Ankle. 1989 Jun;9(6):317-23. doi: 10.1177/107110078900900616. No abstract available. PMID 2663678
- [Result] Davies MS, Weiss GA, Saxby TS. Plantar fasciitis: how successful is surgical intervention? Foot Ankle Int. 1999 Dec;20(12):803-7. doi: 10.1177/107110079902001209. PMID 10609710
- [Result] Pfeffer G, Bacchetti P, Deland J, Lewis A, Anderson R, Davis W, Alvarez R, Brodsky J, Cooper P, Frey C, Herrick R, Myerson M, Sammarco J, Janecki C, Ross S, Bowman M, Smith R. Comparison of custom and prefabricated orthoses in the initial treatment of proximal plantar fasciitis. Foot Ankle Int. 1999 Apr;20(4):214-21. doi: 10.1177/107110079902000402. PMID 10229276
- [Result] Hawke F, Burns J, Radford JA, du Toit V. Custom-made foot orthoses for the treatment of foot pain. Cochrane Database Syst Rev. 2008 Jul 16;2008(3):CD006801. doi: 10.1002/14651858.CD006801.pub2. PMID 18646168
- [Result] Lopez-Lopez D, Rodriguez-Vila I, Losa-Iglesias ME, Rodriguez-Sanz D, Calvo-Lobo C, Romero-Morales C, Becerro-de-Bengoa-Vallejo R. Impact of the quality of life related to foot health in a sample of pregnant women: A case control study. Medicine (Baltimore). 2017 Mar;96(12):e6433. doi: 10.1097/MD.0000000000006433. PMID 28328852
- [Result] Riskowski JL, Hagedorn TJ, Hannan MT. Measures of foot function, foot health, and foot pain: American Academy of Orthopedic Surgeons Lower Limb Outcomes Assessment: Foot and Ankle Module (AAOS-FAM), Bristol Foot Score (BFS), Revised Foot Function Index (FFI-R), Foot Health Status Questionnaire (FHSQ), Manchester Foot Pain and Disability Index (MFPDI), Podiatric Health Questionnaire (PHQ), and Rowan Foot Pain Assessment (ROFPAQ). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S229-39. doi: 10.1002/acr.20554. No abstract available. PMID 22588747
- [Result] Lopez Lopez D, Lopez Martinez NZ, Losa Iglesias ME, Rodriguez Sanz D, Palomo Lopez P, Becerro de Bengoa Vallejo R. Impact on quality of life related to foot health in a sample of menopausal women: a case-control observational study. Climacteric. 2016 Oct;19(5):501-5. doi: 10.1080/13697137.2016.1198314. Epub 2016 Jun 24. PMID 27338169
- [Result] Lopez DL, Callejo Gonzalez L, Losa Iglesias ME, Canosa JL, Sanz DR, Lobo CC, Becerro de Bengoa Vallejo R. Quality of Life Impact Related to Foot Health in a Sample of Older People with Hallux Valgus. Aging Dis. 2016 Jan 2;7(1):45-52. doi: 10.14336/AD.2015.0914. eCollection 2016 Jan. PMID 26816663
- [Result] Grim C, Kramer R, Engelhardt M, John SM, Hotfiel T, Hoppe MW. Effectiveness of Manual Therapy, Customised Foot Orthoses and Combined Therapy in the Management of Plantar Fasciitis-a RCT. Sports (Basel). 2019 May 28;7(6):128. doi: 10.3390/sports7060128. PMID 31141994
- [Result] Rome K, Gray J, Stewart F, Hannant SC, Callaghan D, Hubble J. Evaluating the clinical effectiveness and cost-effectiveness of foot orthoses in the treatment of plantar heel pain: a feasibility study. J Am Podiatr Med Assoc. 2004 May-Jun;94(3):229-38. doi: 10.7547/0940229. PMID 15153583
- [Result] Chuter VH, Searle A, Spink MJ. Flip-flop footwear with a moulded foot-bed for the treatment of foot pain: a randomised controlled trial. BMC Musculoskelet Disord. 2016 Nov 11;17(1):468. doi: 10.1186/s12891-016-1327-x. PMID 27835963